CLINICAL TRIAL: NCT02589860
Title: A Pilot Study: Gene Expression and Bacterial Analysis of Oral Mucositis in Patient's Undergoing Melphalan Conditioning and Autologous Stem Cell Transplant
Brief Title: Analysis of Oral Mucositis in Patient's Undergoing Melphalan Conditioning and Autologous Stem Cell Transplant
Status: Withdrawn | Type: Observational
Why Stopped: No accrual
Sponsor: Sherif S. Farag (Other)
Responsible Party: Sponsor-Investigator, Sherif S. Farag, Professor of Medicine and Medical and Molecular Genetics, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: IUSCC-0536
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Mucositis; Multiple Myeloma; Amyloidosis; Oral Mucositis
Keywords: Stem Cell Transplantation
MeSH Terms: conditions — Mucositis; Multiple Myeloma; Amyloidosis; Stomatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cells collected from oral mucosal samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Melphalan kinetic study — Concentration of Melphalan in plasma samples
Genetic: Oral bacterial study — DNA from oral buccal mucosal cells will be sequenced for bacterial composition
Genetic: Gene expression study — RNA from oral buccal mucosal cells will be analyzed to compare gene expression

SUMMARY:
This is a pilot study to explore and identify changes in molecular processes within the oral mucosa that are associated with the development of oral mucositis (OM) in patients treated with Melphalan who undergo autologous peripheral blood stem cell transplantation.

DETAILED DESCRIPTION:
This is an exploratory observational (non-therapeutic) study to collect blood and buccal mucosal samples to evaluate RNA expression, assess bacterial colonization, and plasma Melphalan concentrations in approximately 50 eligible patients.

All study samples will be collected from participants while they are hospitalized to receive standard of care high-dose Melphalan (HDM) chemotherapy and autologous peripheral blood stem cell transplantation (ASCT). Patients who receive this treatment are typically admitted the day before HDM. The day after HDM, patients receive ASCT and remain hospitalized for approximately 21 days, or until their absolute neutrophil count increases to at least 500 cells per mm3 and they are no longer considered neutropenic.

Patients will have blood samples collected for pharmacokinetic analysis at approximately 0 minutes (before infusion begins), 15 minutes (during the infusion), 30 minutes (at the end of infusion), 60 minutes, 90 minutes, 120 minutes, and 180 minutes after the start of Melphalan infusion.

A buccal swab will be done to collect mucosal bacterial samples using paper strips (Periopaper) or a sterile cotton tipped swab brushed against the right and left buccal mucosa for approximately 15-30 seconds at the following time points:

1. Within 24 hours PRIOR to administration of Melphalan
2. Day +3 AFTER transplantation
3. Upon development of OM (approximately on days +7-10)
4. Upon recovery of absolute neutrophil count (ANC) to greater than 500/mm3, or on discharge, whichever occurs first, in patients who developed OM

A buccal scraping will be done for gene expression using a dermatologic curette taken from the right and left buccal mucosa at the following time points:

1. Within 24 hours PRIOR to administration of Melphalan
2. Day +3 AFTER transplantation Note: Patients' mouths will be rinsed with Mary's Magic mouthwash prior to the procedure for 15 seconds, which will allow for removal of food particles, colonized bacteria and anesthetization of oral mucosa. During procedure, any signs of patient discomfort will be monitored. If patient expresses discomfort, additional oral topical anesthetic will be utilized to de-sensitive buccal mucosa.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple myeloma (MM) or systemic light-chain amyloidosis who are receiving high-dose Melphalan (HDM) and autologous peripheral blood stem cell transplantation (ASCT).
2. Age is greater than 18 years old
3. Patients receiving a total Melphalan dose of 140-200 mg/m2 as the preparative regimen
4. No prior history of allogeneic stem cell transplantation
5. Patients otherwise meeting all standard institutional criteria for ASCT

Exclusion Criteria:

1. Patients who do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Melphalan who undergo autologous stem cell transplant at the Indiana University Health Melvin and Bren Simon Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Gene expression | 30 days
  RNA sequencing from oral buccal mucosal cells
Bacterial colonization | 30 days
  DNA sequencing of bacteria in oral buccal mucosal cells
Melphalan exposure | 30 days
  Concentration of Melphalan in plasma samples

CONTACTS AND LOCATIONS:
Overall Officials: Sheriff Farag, M.D., Ph.D., Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (2):
- United States (2):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana